CLINICAL TRIAL: NCT03159338
Title: The Effect of Platelet-rich Fibrin on Nerve Regeneration After Bilateral Sagittal Split Osteotomy of the Mandible
Brief Title: Platelet-rich Fibrin on Nerve Regeneration After Bilateral Sagittal Split Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, Assistant professor of oral and maxillofacial surgery, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 30345
Record Dates: First submitted 2017-05-02; First posted 2017-05-18 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Paresthesia; Anesthesia, Local; Neurosensory Disorder
MeSH Terms: conditions — Paresthesia; Sensation Disorders

STUDY DESIGN:
Intervention Model Description: one side of osteotomies randomally will be considered as a treatment group and another side as a control group.
Who Masked: Participant
Masking Description: Investigator will be blunt about side of treatmen and control.None of surgical team will be as an investigator.Patients will unware about which side is treatment or control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): One side of osteotomies will be considered as a treatment arm (randomly) which Platelet rich fibrin will be used with rigid fixation
  Interventions: Biological: Platelet rich fibrin
- Control group (Placebo Comparator): In control site , placebo gel will be placed before rigid fixation
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Platelet rich fibrin — Platelet rich fibrin will be prepared by taking 20 cc blood and centrifugation with 28000 rpm.
  Arms: treatment group
Biological: Placebo — In control group , after spliting the osteotomy site before fixation a placebo gel will be placed
  Arms: Control group

SUMMARY:
Patients who have mandibular deformity and will undergo bilateral sagittal split osteotomy will be included in the study.One side of the osteotomies randomly will be considered as study group and another side as a control group.In the study group , platelet rich fibrin will be placed after osteotomy and before rigid fixation.In the control group, fixation will be done without Platelet-rich Fibrin (PRF).Neurosensory disturbance will be evaluated 6 and 12 months after surgeries.

DETAILED DESCRIPTION:
Patients who have mandibular deformity and will undergo bilateral sagittal split osteotomy will be included in the study.One side of the osteotomies randomly will be considered as study group and another side as a control group.In the study group , platelet rich fibrin will be placed after osteotomy and before rigid fixation.In the control group fixation will be done without Platelet-rich Fibrin. Before starting the surgical procedure, 20 mL of venous blood will take and placed in a centrifuge for 12 minutes with 28000rpm. After centrifugation, the cap will be removed from each tube and they will be placed into a sterile rack L-PRF™. Fibrin matrix will prepare. The L-PRF™ will be removed from the tube. Then, the clot right beneath the red blood cell clot will be placed on the surface tray and covered. Five minutes will be waited before removing and using the fibrin matrix.Neurosensory disturbance will be evaluated in 6 and 12 months after osteotomies by two-point discrimination (TPD) test and pin tactile discrimination(PTD) tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have class II or III deformity and will undergo bilateral sagittal split osteotomy

Exclusion Criteria:

* Patients who have bad split or obvious nerve injury during surgery will be removed from study inclusion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Two-point discrimination (TPD) test | TPD will be assessed after 6 months
  Two point discrimination will be measured based on the distance of two points (mm)
Two-point discrimination | Two-point discrimination will be evaluated after12 months intervals
  Two point discrimination will be measured based on the distance of two points (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Tabrizi, DMD, Principal Investigator — Shiraz University of Medical Sciences
Locations (2):
- Iran (2):
  - Shiraz university of medical sciences, Shiraz
  - Taleghani Hospital, Tehran

IPD SHARING:
Plan to Share IPD: Undecided